CLINICAL TRIAL: NCT01540539
Title: Intravenous/Subcutaneous FIH Study of REGN1154 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: R1154-HV-1116
Record Dates: First submitted 2012-02-23; First posted 2012-02-28 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Dosing cohort 1 (Experimental)
  Interventions: Drug: REGN1154 or placebo
- Dosing cohort 2 (Experimental)
  Interventions: Drug: REGN1154 or placebo
- Dosing cohort 3 (Experimental)
  Interventions: Drug: REGN1154 or placebo
- Dosing cohort 4 (Experimental)
  Interventions: Drug: REGN1154 or placebo
- Dosing cohort 5 (Experimental)
  Interventions: Drug: REGN1154 or placebo
- Dosing cohort 6 (Experimental)
  Interventions: Drug: REGN1154 or placebo
- Dosing cohort 7 (Experimental)
  Interventions: Drug: REGN1154 or placebo
- Dosing cohort 8 (Experimental)
  Interventions: Drug: REGN1154 or placebo

INTERVENTIONS:
Drug: REGN1154 or placebo — Participants will receive active drug or placebo

SUMMARY:
The purpose of this study is to study the safety and tolerability of intravenous (IV) and subcutaneous (SC) administration of REGN1154 in normal healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women between the ages of 18 and 65; women must be postmenopausal or surgically sterile
2. Body mass index (BMI) between 18.0 and 30.0 kg/m2, inclusive
3. Willing, committed, and able to return for ALL clinic visits and complete all study-related procedures
4. Able to read or to understand the consent process, and willing to sign the informed consent form (ICF)

Exclusion Criteria:

Exclusion criteria include, but are not limited to the following:

1. Any illness or condition that would adversely affect the subject's participation in this study
2. Any clinically significant abnormalities observed during the screening visit
3. Use of certain medications taken before the screening visit
4. Onset of a new exercise routine or major change to a previous exercise routine within 4 weeks prior to screening visit
5. Hospitalization within 60 days of the screening visit
6. Any condition that would place the subject at risk, interfere with participation in the study
7. History of or positive human immunodeficiency virus (HIV) screen result at the screening visit
8. History of certain other conditions
9. Positive urine, drug or alcohol screen result at screening
10. Known sensitivity to any of the components of the investigational product formulation
11. Participation in any clinical research study evaluating another investigational drug or therapy within 30 days or at least 5 half-lives (whichever is longer), of the investigational drug prior to the screening visit
12. Live/attenuated vaccinations within 12 weeks of screening or during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Total number and severity of TEAEs | Day 1 through Day 113
  TEAEs (Treatment-emergent adverse events)

SECONDARY OUTCOMES:
Serum concentration | Day 1 through Day 113
  Serum concentrations of REGN1154 over time
Presence or absence of antibodies | Day 1 through Day 113
  Presence or absence of antibodies against REGN1154 over time.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Melbourne, Australia